CLINICAL TRIAL: NCT04182074
Title: A Prospective Registry-based Cohort Study to Monitor the Diagnosis and Management of Acute Leukaemia in Pregnancy.
Brief Title: Monitoring the Diagnosis and Management of Acute Leukaemia In Pregnancy Study.
Acronym: LIPS
Status: Completed | Type: Observational
Sponsor: University of Hull (Other)
Responsible Party: Sponsor
Other Study IDs: UoH 2019/01
Record Dates: First submitted 2019-11-20; First posted 2019-12-02 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Acute Leukemia
Keywords: Pregnancy; Treatment; Diagnosis; Delivery
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute leukaemia (AL) is an aggressive but potentially curable cancer that can affect women of childbearing age. When a pregnancy is complicated by a diagnosis of AL, clinicians face a complex dilemma: to balance risking the mother's survival through delaying treatment, against the potential harm to the foetus through exposure to cancer drugs. Reports suggest that, providing the first trimester is avoided, successful treatment of AL during pregnancy is possible, and considered safe. However, there is currently no standard approach to treatment of these women.

This observational study aims to monitor and record the current treatment and outcomes of patients diagnosed with acute leukaemia during or prior to pregnancy. Patients will receive the treatment recommended by their doctor, the study will not alter the treatment pathway of participants. This study will establish a new research database of Leukaemia in Pregnancy, initially collecting data from cases since August 2009, and any new cases that are diagnosed during the current funding period.

The initial planned analyses from this dataset will enable more robust, evidence-based recommendations to be made on how to monitor and manage these patients, and will add value to and improve the existing British Committee for Standards in Haematology (BCSH) guidelines, which were largely derived from expert opinion. This should enable healthcare professionals to have greater confidence in managing these patients, leading to a more standardised approach to providing high quality care. The study will benefit National Health Service (NHS) Trusts and patients across the United Kingdom (UK) through more informed clinical decision making with regards to the care they receive. It will also provide an important data resource which researchers can apply to use in further analyses, with plans to continue data collection if further funding is obtained.

DETAILED DESCRIPTION:
A registry-based cohort study to identify and collect data on all women receiving a diagnosis of AL or high-risk myelodysplastic syndrome (MDS), and all women with a history of AL or high-risk MDS who fall pregnant within the study period. This is an observational study, and patients will receive usual care as determined by their Loco-regional multidisciplinary team.

We aim to approach all consultant haematologists involved in the care of a woman diagnosed with AL during pregnancy, and request that they report all known cases, creating a national dataset. For prospective cases, women will be identified at diagnosis and tracked throughout their pregnancy to allow comparison of the respective outcomes for both mother and neonate. There will be additional follow-up points at 2 and 4 years, to accurately document the subsequent outcomes of the mother and obtain details of any further pregnancies they may have had. The follow-up periods were chosen as two and four years. Two years is where the most incidences of relapse occur, and four years is considered decisive with regards to remission. In addition, consultant haematologists across the UK will be asked to provide retrospective data on any cases occurring since August 2009 (both pre-and post-introduction of the 2015 BCSH guidelines), to gain an overview of current and past approaches to patient management, and to serve as comparators to assess the current and future impact of the BCSH guidelines.

Consent will be sought from the patient whenever reasonably practicable for the use of the information in the database. In historic cases when to patient is no longer in contact with the hospital (e.g. no longer in clinical follow-up), to avoid causing any emotional distress the relevant approvals will be gained to process these cases without consent. All information will be retrieved from the patient's medical records and will require no further patient involvement beyond consenting for the use of their information.

Data from the LIPS database will be hosted and managed by the Hull Health Trials Unit (HHTU) using their secure online data capture system RedCap Cloud (RCC) and BOX Governance file storage system. HHTU hold a NHS Digital Data Security and Protection Toolkit covering these information systems. RCC is a cloud based electronic data collection system provided by nPhase. Data is stored on dedicated RCC hardware in European Union data centres (including real-time backup) managed by Amazon Web Services to industry standards outlined in ISO 27001, PCI DSS, SOC 1 -3, FISMA, CIS, CSA, NIST and UK Cloud Security Principles. Data is encrypted at rest and in transit. RCC deliver compliance to HIPAA, CFR Part 11, and EMEA Annex 11.

Data checks are built in to the database to compare inputted data with predefined ranges and values with data management according to the data management plan with data querying of any missing or anomalous data. A statistical analysis plan will be prepared before the analysis of the initial dataset.

ELIGIBILITY:
Inclusion Criteria:

* Women who have a diagnosis of acute leukaemia (AL) or high-risk myelodysplasia (MDS) in pregnancy, or who have later conceived after receiving previous treatment for either AL or high-risk MDS.

Exclusion Criteria:

* Pregnant women not meeting the inclusion criterion.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Secondary care in the UK
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of deaths and complications during pregnancy and up to one month after delivery. | Up to 1 month after delivery.
  Morbidity and mortality outcomes of women treated for AL or high-risk MDS during pregnancy.
Number of neonatal deaths and complications during pregnancy and up to one month after delivery. | Up to 1 month after delivery.
  Short term morbidity and mortality outcomes for neonates born by women who were treated for AL or high-risk MDS during pregnancy.
Number of deaths and complications during pregnancy. | Up to 1 month after delivery.
  Morbidity and mortality outcomes during pregnancy of women previously treated for AL or high-risk MDS.
Number of neonatal deaths and complications during pregnancy and up to one month after. | Up to 1 month after delivery.
  Short term morbidity and mortality outcomes of neonates born by women who were previously treated for AL or high-risk MDS.

SECONDARY OUTCOMES:
Number and types of treatments used during the pregnancy. | Up to the 9 months of the pregnancy.
  Current treatment practices for women diagnosed with AL or high-risk MDS during pregnancy.
Number and types of monitoring procedures used during the pregnancy. | Up to the 9 months of the pregnancy.
  Current monitoring practices for women diagnosed with AL or high-risk MDS during pregnancy.
Number and types of treatments who subsequently become pregnant. | Up to the 9 months of the pregnancy.
  Current treatment practices for women who became pregnant after previously receiving therapy for AL or high-risk MDS.
Number and types of monitoring procedures used during the pregnancy in women who previously received therapy for AL or high-risk MDS. | Up to the 9 months of the pregnancy.
  Current monitoring practices for women who became pregnant after previously receiving therapy for AL or high-risk MDS.
Number of deaths during the follow-up period. | Mother - Up to 4 years after delivery.
  Long term mortality of the woman.
Number of further pregnancies and outcome of the pregnancy. | Mother - Up to 4 years after delivery.
  Long term treatment effects on the fertility.
Number of women with treatment-related adverse events as assessed by CTCAE v4.0. | Mother - Up to 4 years after delivery.
  Long term side effect of treatment to the woman.
Number of congenital abnormalities reported in the infant up to 28 days after delivery | Child - Up to 28 days after birth.
  Side effects of treatment to the infant.

CONTACTS AND LOCATIONS:
Overall Officials: Sahra Ali, MBChB, MRCP, FRCPath, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; David Allsup, Principal Investigator — Hull York Medical School
Locations (1):
- Hull University Teaching Hospital NHS Trust, Hull, United Kingdom

REFERENCES:
- [Background] Ali S, Jones GL, Culligan DJ, Marsden PJ, Russell N, Embleton ND, Craddock C; British Committee for Standards in Haematology. Guidelines for the diagnosis and management of acute myeloid leukaemia in pregnancy. Br J Haematol. 2015 Aug;170(4):487-95. doi: 10.1111/bjh.13554. Epub 2015 Jun 17. PMID 26081614
- [Background] Northgraves M, Allsup D, Cohen J, Huang C, Turgoose J, Ali S. A prospective registry-based cohort study of the diagnosis and management of acute leukaemia in pregnancy: Study protocol. PLoS One. 2022 Feb 7;17(2):e0263195. doi: 10.1371/journal.pone.0263195. eCollection 2022. PMID 35130292